CLINICAL TRIAL: NCT06365931
Title: Physiological and Functional Effects of Percutaneous Neuromodulation vs Transcutaneous Neuromodulation in the Clubfoot Approach in Post-stroke Patients. Clinical Trial
Brief Title: Physiological and Functional Effects of Percutaneous Neuromodulation vs Transcutaneous Neuromodulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Alejandro Caña Pino, Clinical Proffesor, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 160224
Record Dates: First submitted 2024-04-03; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Stroke/Brain Attack
Keywords: Neuromodulation; clubfoot; percutaneous; transcutaneous; tibialis anterior
MeSH Terms: conditions — Stroke; Clubfoot | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- G1 (percutaneous neuromodulation) (Experimental): Patients will receive a needle circuit approaching the deep peroneal nerve in an ultrasound-guided manner. They will receive a symmetrical biphasic current of 20-30Hz and 250 μs at tolerable intensity.
  Interventions: Device: Percutaneous neuromodulation; Device: Percutaneous neuromodulation or Transcutaneous neuromodulation (optional)
- G2 (transcutaneous neuromodulation) (Experimental): Patients will have a superficial electrode circuit placed over the belly of the tibialis anterior muscle. They will receive a symmetrical biphasic current of 20-30Hz and 250 μs at tolerable intensity.
  Interventions: Device: Transcutaneous neuromodulation; Device: Percutaneous neuromodulation or Transcutaneous neuromodulation (optional)
- G3 (placebo-percutaneous group) (Placebo Comparator): Patients will receive the neuromodulation circuit with needles at 0 intensity, approaching the deep peroneal nerve in an ultrasound-guided manner
  Interventions: Device: Placebo-percutaneous; Device: Percutaneous neuromodulation or Transcutaneous neuromodulation (optional)
- G4 (placebo-transcutaneous group) (Placebo Comparator): Patients will have the electrodes placed over the tibialis anterior muscle at intensity 0.
  Interventions: Device: Placebo-transcutaneous; Device: Percutaneous neuromodulation or Transcutaneous neuromodulation (optional)

INTERVENTIONS:
Device: Percutaneous neuromodulation — Patients will receive a needle circuit approaching the deep peroneal nerve in an echoguided manner. They will receive a symmetrical biphasic current of 20-30Hz and 250 μs at tolerable intensity.
  Arms: G1 (percutaneous neuromodulation)
Device: Transcutaneous neuromodulation — Patients will have a superficial electrode circuit placed over the belly of the tibialis anterior muscle. They will receive a symmetrical biphasic current of 20-30Hz and 250 μs at tolerable intensity.
  Arms: G2 (transcutaneous neuromodulation)
Device: Placebo-percutaneous — Patients will have the neuromodulation circuit placed with needles at 0 intensity, approaching the deep peroneal nerve in an ultrasound-guided manner.
  Arms: G3 (placebo-percutaneous group)
Device: Placebo-transcutaneous — patients will have the electrodes placed over the tibialis anterior muscle at intensity 0.
  Arms: G4 (placebo-transcutaneous group)
Device: Percutaneous neuromodulation or Transcutaneous neuromodulation (optional) — Study participants who wish to continue may be randomized to receive a 10-session intervention program. The intervention to be received will consist of 10 sessions of percutaneous neuromodulation or 10 sessions of transcutaneous neuromodulation, two sessions per week.

SUMMARY:
INTRODUCTION: Clubfoot, drop foot or clubfoot, is a disorder that prevents reaching 100º of dorsiflexion actively. Its etiology is varied, and may be due to congenital problems, direct alteration of the bone structure, spasticity or shortening of the posterior musculature (triceps suralis), a neurological factor or a combination of several. Thus, we can differentiate between congenital clubfoot and acquired clubfoot. Stroke is one of the main causes of acquired clubfoot, which is due to paralysis of the dorsiflexor musculature and/or spasticity of the plantar flexor musculature. Electrical stimulation is able to increase muscle activation by depolarization of the motor plate and modulation of nerve conduction. This can be done transcutaneously, through surface electrodes or percutaneously through needles, so neuromodulation is presented as a tool applicable to the pathology of the equine foot, if we take into account the increased activation of the dorsiflexors of the foot.

OBJECTIVE: The main objective is to evaluate which of the techniques, percutaneous or transcutaneous, is more effective for the approach of clubfoot in post-stroke patients.

METHODOLOGY: a clinical trial with randomized probabilistic assignment in four groups is proposed: G1 (percutaneous neuromodulation): patients will receive a needle circuit approaching the deep peroneal nerve in an ultrasound-guided manner. They will receive a 20-30Hz symmetrical biphasic current; G2 (transcutaneous neuromodulation): patients will have a superficial electrode circuit placed over the belly of the tibialis anterior muscle. They will receive a symmetrical biphasic current of 20-30Hz; G3 (placebo-percutaneous group): in which the patients will receive the neuromodulation circuit with needles at 0 intensity; G2 (placebo-transcutaneous group): the patients will receive the electrodes at 0 intensity over the belly of the tibialis anterior muscle.

The variables to be analyzed are: anthropometric variables (age, weight, height, BMI), muscle oxygenation (SatO2, O2Hb, HHb and THb), muscle strength of the foot dorsiflexors measured with dynamometer, muscle activation by surface electromyography, active and passive joint balance with goniometry or inclinometer, assessment of gait and balance, assessment of load distribution by static and dynamic pressure platform, spasticity and questionnaire on quality of life and functionality. The acute effects after one intervention session (pre-post intervention of one session) and the effects after a 10-session program will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old.
* Have had a stroke or brain damage acquired at least 1 year ago.
* Have a muscle balance in the dorsiflexor musculature of the foot less than or equal to 3/5 on the Daniels scale.

Exclusion Criteria:

* Contraindication to electrotherapy.
* Needle phobia or panic (in the case of having been assigned to the percutaneous group).
* Severe cognitive impairment that prevents collaboration in the performance of the activity.
* Failure to meet the inclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Muscle activity | 1 day
  MDurance surface electromyography
Displacement of the center of pressures (CoP) | 1 day
  Postural stability: baropodometric platform
Articular amplitude | 1 day
  Dorsal flexion using goniometer
Balance | 1 day
  Timed Up and Go (TUG)
Balance | 1 day
  Tinetti scale: The test is divided into two parts, the assessment of balance on the one hand and gait on the other. To do this we will ask the patient different movements and activities that we will score from 0 to 2, depending on the section, being the maximum score in the balance 16 points and 12 points in the gait.
Gait | 1 day
  10 minutes walking test
Tissue oxygen in muscle | 1 day
  Oximeter. Moxy-3 in the thigh
Muscular strength | 1 day
  Tibialis anterior strength by dynamometry
Functionality | 1 day
  ECVI-38 scale (Quality of Life Scale for Stroke): 38 items hypothetically grouped into eight domains: physical state, communication, cognition, emotions, feelings, basic activities of daily living, common activities of daily living, and socio-familial functions.; plus two additional questions on sexual function and work activity.
quality of life index | 1 day
  ECVI-38 scale (Quality of Life Scale for Stroke): 38 items hypothetically grouped into eight domains: physical state, communication, cognition, emotions, feelings, basic activities of daily living, common activities of daily living, and socio-familial functions.; plus two additional questions on sexual function and work activity.
Spasticity | 1 day
  Ashworth scale: scale from 0 to 4. 0 means mild muscle tone and 4 means high hypertonicity.

CONTACTS AND LOCATIONS:
Locations (1):
- Mª Dolores Apolo Arenas, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No